CLINICAL TRIAL: NCT00041756
Title: Efficacy and Safety of PG-530742 in the Treatment of Mild to Moderate Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001065
Record Dates: First submitted 2002-07-16; First posted 2002-07-17 (Estimated); Results first posted 2011-11-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Primary Disease: Knee Primary Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo
- 25 mg PG-530742 (Experimental): 25 mg PG-530742
  Interventions: Drug: PG-530742
- 50 mg PG-530742 (Experimental): 50 mg PG-530742
  Interventions: Drug: 50 mg PG-530742
- 100 mg PG-530742 (Experimental): 100 mg PG-530742
  Interventions: Drug: 100 mg PG-530742
- 200 mg PG-530742 (Experimental): 200 mg PG-530742
  Interventions: Drug: 200 mg PG-530742

INTERVENTIONS:
Drug: PG-530742 — One 25 mg PG-530742 tablet, twice daily for for one year
  Arms: 25 mg PG-530742
Drug: Placebo — One placebo tablet, twice daily for for one year
  Arms: Placebo
Drug: 50 mg PG-530742 — One 50 mg PG-530742 tablet, twice daily for for one year
  Arms: 50 mg PG-530742
Drug: 100 mg PG-530742 — 100 mg PG-530742 tablet, twice a day for one year
  Arms: 100 mg PG-530742
Drug: 200 mg PG-530742 — 200 mg PG-530742 tablet, twice a day for one year
  Arms: 200 mg PG-530742

SUMMARY:
Matrix metalloproteinases (MMPs) have been implicated in the cartilage degradation. PG-530742 inhibits some MMPs, potentially limiting cartilage degradation and disease progression. This study will test the efficacy and safety of PG-530742 in the treatment of mild to moderate knee osteoarthritis.

DETAILED DESCRIPTION:
Matrix metalloproteinases have been implicated in the cartilage degradation that occurs in osteoarthritis. PG-530742 inhibits some of these matrix metalloproteinases, thus potentially limiting cartilage degradation and disease progression. This study will test the efficacy and safety of PG-530742 in the treatment of mild to moderate knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate knee osteoarthritis confirmed by a radiographic technique.

Exclusion Criteria:

* secondary knee osteoarthritis;
* diseases other than osteoarthritis that could cause knee pain;
* any disease or intervention (surgery, intra-articular injection) that would have an impact on knee pain or mobility;
* drugs that act potentially on the bone or cartilage component of the knee joint.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2002-07; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Beary, MD, Study Director — Procter and Gamble
Locations (23):
- Hungary (7):
  - Rehabilitation Hospital, Gizella telep, Visegrád, Gizella Telep
  - Petz A. Country Hospital, Department of Rheumatology, Hid utca 2., Győr, Hid Utica 2
  - National Institute of Rheumatology and Physiotherapy, Dept. of Rheumatology and Immunology, Frankel Leo u. 38-40, Budapest
  - National Institute of Rheumatology and Physiotherapy, Dept. of Rheumatology I and Metabolic Osteology, Frankel Leo u. 38-40, Budapest
  - National Institute of Rheumatology and Physiotherapy, Dept. of Rheumatology IV., Frankel Leo u. 38-40, Budapest
  - Orthopedic Clinic, Karolina ut 17, Budapest
  - Szent Ferenc Hospital, Department of Rheumatology, Csabai Kapu 42., Miskolc
- United Kingdom (16):
  - 95 Stanwell Road, Ashford, Middlesex
  - Royal National Orthapaedic Hsopital, Brackley Hill, Stanmore, Middlesex
  - St Thomas Hospital, Lambeth Place Road, London, Se17eh
  - The Crouch Oak Practice, 45 Station Road, Addlestone, Addlestone, Surrey
  - The Medical Centre, Kingston Avenue, East Horsley, Surrey
  - Bridge House Medical Centre, Scholars Lane, Stratford-upon-Avon, Warwickshire
  - Pound Hill Surgery, 1 Crawley Lane, Pound Hill, Crawley, West Sussex
  - Dept of Rheumatology Selly Oak Hospital, Raddleburn Road, Selly Oak, Birmingham
  - Synexus Birmingham Clinical Research Centre, Birmingham Research Park, Edgbaston
  - Grosvenor Medical Centre Clinical Trials Unit, 18 upper Grosvenor Road, Tunbridge Wells, Kent
  - Dept of Rheumatology Whipps Cross University Hospital, Whipps Cross Road, London
  - Dept of Rheumatology Dulwich Hospital, East Dulwich, London
  - Rheumatology Department, Fourth Floor, Thomas Guy House, St Guy's House, London Bridge
  - Synexus Reading Clinical Research Centre, Whiteley Glebe, 11 Glebe Road, off Christchurch Gardens, Reading
  - Hildenborough Medical Group, Trenchwood Surgery, 264 Shipbourne Road, Tonbridge
  - Synexus Wrightington, Wrightington Hospital, Hall Lane, Awpley Bridge, Wigan

REFERENCES:
- [Derived] Krzeski P, Buckland-Wright C, Balint G, Cline GA, Stoner K, Lyon R, Beary J, Aronstein WS, Spector TD. Development of musculoskeletal toxicity without clear benefit after administration of PG-116800, a matrix metalloproteinase inhibitor, to patients with knee osteoarthritis: a randomized, 12-month, double-blind, placebo-controlled study. Arthritis Res Ther. 2007;9(5):R109. doi: 10.1186/ar2315. PMID 17958901

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Tablet: Placebo tablet dosed BID
- 25 mg PG-530742: 25 mg PG-530742 dosed BID
- 50 mg PG-530742: 50 mg PG-530742 dosed BID
- 100 mg PG-530742: 100 mg PG-530742 dosed BID
- 200 mg PG-530742: 200 mg PG-530742 dosed BID
Period: Overall Study
Arm/Group | Placebo Tablet | 25 mg PG-530742 | 50 mg PG-530742 | 100 mg PG-530742 | 200 mg PG-530742
Started | 77 | 80 | 79 | 80 | 79
Completed | 69 | 65 | 66 | 64 | 19
Not Completed | 8 | 15 | 13 | 16 | 60
Not completed — Adverse Event | 4 | 10 | 6 | 11 | 34
Not completed — Protocol Violation | 1 | 1 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 3 | 3 | 4 | 2 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0
Not completed — Unable to meet protocol criteria | 0 | 0 | 1 | 0 | 1
Not completed — Data Monitoring Committee Recommendation | 0 | 0 | 0 | 0 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Tablet | 25 mg PG-530742 | 50 mg PG-530742 | 100 mg PG-530742 | 200 mg PG-530742 | Total
Number analyzed (Participants) | 77 | 80 | 79 | 80 | 79 | 395
Age Continuous [Mean (Standard Deviation); unit: years] | 62.0 (0.92) | 62.4 (0.86) | 62.6 (0.92) | 62.9 (0.95) | 63.1 (0.80) | 62.6 (0.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 60 | 61 | 57 | 49 | 281
  Male | 23 | 20 | 18 | 23 | 30 | 114
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian | 0 | 0 | 0 | 0 | 0 | 0
  Asian Oriental | 0 | 0 | 0 | 0 | 0 | 0
  Black | 0 | 1 | 1 | 1 | 0 | 3
  Caucasian | 77 | 79 | 77 | 75 | 76 | 384
  Hispanic | 0 | 0 | 0 | 0 | 0 | 0
  Asian Indian | 0 | 0 | 1 | 4 | 3 | 8
  Multi-Racial | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Minimum Joint Space Width in the Medial Compartment of the Tibiofemoral Joint of the Signal Knee After 1 Year of Treatment
Description: The structural primary efficacy endpoint is the 1-year change from baseline in minimum joint space width (JSW) in the medial compartment of the tibiofemoral joint of the signal knee, as measured by microfocal knee radiographs obtained in the semi-flexed position.
Time Frame: baseline and 12 months
Population: An intent-to-treat (ITT) analysis was conducted on all patients who were randomized and took at least one dose of study drug. Any missing data for these patients was not imputed in the primary analysis.
  analysis.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo Tablet | 25 mg PG-530742 | 50 mg PG-530742 | 100 mg PG-530742 | 200 mg PG-530742
Number analyzed (Participants) | 71 | 66 | 67 | 69 | 52
mm | -0.1361 (0.0627) | -0.0442 (0.0624) | -0.2261 (0.0650) | -0.2000 (0.0650) | -0.1916 (0.0723)

2. Primary Outcome: Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Total Score at 1 Year
Description: The symptomatic primary efficacy endpoint is the change in total WOMAC scores after 1 year of treatment. The WOMAC consists of 24 items divided into 3 subscales: Pain (5 items), Stiffness (2 items), Physical Function (17 items). The WOMAC uses descriptors for all items: none, mild moderate, severe, and extreme (corresponding to an ordinal scale of 0-4.) Scores are summed for items in each subscale, with possible ranges as follows: pain=0-20, stiffness=0-8, physical function=0-68. The total WOMAC score is created by summing the items for all three subscales (min=0, max=96)
Time Frame: baseline and 12 months
Population: An intent-to-treat (ITT) analysis was conducted on all patients who were randomized and took at least one dose of study drug. Any missing data for these patients was not imputed in the primary analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo Tablet | 25 mg PG-530742 | 50 mg PG-530742 | 100 mg PG-530742 | 200 mg PG-530742
Number analyzed (Participants) | 67 | 61 | 62 | 62 | 30
Scores on a scale | -9.1 (2.81) | -6.7 (2.78) | -10.0 (2.88) | -5.8 (2.92) | -9.3 (3.96)

ADVERSE EVENTS:
Arm/Group | Placebo Tablet | 25 mg PG-530742 | 50 mg PG-530742 | 100 mg PG-530742 | 200 mg PG-530742
Serious Adverse Events (participants affected / at risk) | 8/77 | 7/80 | 12/79 | 10/80 | 17/79
Other Adverse Events (participants affected / at risk) | 37/77 | 41/80 | 34/79 | 43/80 | 44/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Tablet (N=77) | 25 mg PG-530742 (N=80) | 50 mg PG-530742 (N=79) | 100 mg PG-530742 (N=80) | 200 mg PG-530742 (N=79)
Athralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 4 (4) | 3 (3)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pneumonia NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure NOS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaemia NOS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atioventricular block NOS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia NOS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract unilateral (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal erosions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric erosions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibrosis NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biopsy lymph gland abnormal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia NOS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periostitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toe deformities NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc herniation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dupuytren's contracture (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibrositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spondylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertegrobasilar insufficiency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure NOS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral stricture (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatic hypertrophy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage NOS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension NOS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Tablet (N=77) | 25 mg PG-530742 (N=80) | 50 mg PG-530742 (N=79) | 100 mg PG-530742 (N=80) | 200 mg PG-530742 (N=79)
Blood and lymphatic system disorders (Overall) (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 3 (3)
Cardiac disorders (Overall) (Cardiac disorders) | 1 (1) | 4 (6) | 8 (8) | 7 (10) | 4 (5)
Ear and labyrinth disorders (Overall) (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Eye disorders (Overall) (Eye disorders) | 3 (6) | 3 (4) | 5 (6) | 2 (2) | 3 (3)
Gastrointestinal disorders (Overall) (Gastrointestinal disorders) | 14 (31) | 14 (21) | 15 (25) | 16 (34) | 19 (37)
General disorders and administration site conditions (Overall) (General disorders) | 5 (7) | 11 (14) | 12 (13) | 9 (11) | 19 (20)
Infections and infestation (Overall) (Infections and infestations) | 22 (37) | 26 (40) | 16 (18) | 24 (35) | 16 (22)
Injury, poisoning and procedural complications (Overall) (Injury, poisoning and procedural complications) | 6 (9) | 4 (4) | 6 (7) | 7 (7) | 5 (5)
Investigations (Overall) (Investigations) | 9 (14) | 16 (31) | 12 (19) | 9 (16) | 10 (23)
Metabolism and nutrition disorders (Overall) (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 3 (4) | 2 (2)
Musculoskeletal and connective tissue disorders (Overall) (Musculoskeletal and connective tissue disorders) | 37 (91) | 41 (104) | 34 (85) | 43 (135) | 44 (154)
Neoplasms benign, malignant and unspecified (Overall) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 4 (4) | 2 (3) | 0 (0)
Nervous system disorders (Overall) (Nervous system disorders) | 7 (8) | 12 (16) | 10 (15) | 7 (7) | 7 (10)
Psychiatric disorders (Nervous system disorders) | 4 (4) | 2 (3) | 3 (4) | 1 (1) | 4 (6)
Renal and urinary disorders (Renal and urinary disorders) | 4 (4) | 1 (1) | 2 (2) | 3 (3) | 5 (5)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 10 (12) | 6 (8) | 7 (13) | 7 (8)
Skin and subcutaneous tissue disorders (Overall) (Skin and subcutaneous tissue disorders) | 7 (9) | 8 (9) | 8 (10) | 2 (3) | 2 (2)
Vascular disorders (Vascular disorders) | 8 (9) | 7 (7) | 3 (3) | 6 (7) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other